CLINICAL TRIAL: NCT01214512
Title: Performance Evaluation of the Micromedic CD24 Western Blot and ELISA in Vitro Diagnostic Assay
Brief Title: Performance Evaluation of the Micromedic CD24 in Vitro Diagnostic Assay
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MMC10097/2010k-CTIL
Record Dates: First submitted 2010-09-14; First posted 2010-10-05 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-03

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fresh blood samples are collected and separated. Plasma is collected and stored and rest is discarded of. Leukocytes are separated, lysed and the supernatant is stored. As DNA is retained in the pellet, which is discarded, no DNA is retained in the samples stored.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: blood-sample based diagnostic assay — A blood sample will be used in a Western blot and ELISA assay to determine CD24 levels

SUMMARY:
This study is aimed to evaluate the performance of the Micromedic CD24 assay in identifying colorectal adenoma using Western blot and ELISA assays. These assays are designed to detect CD24 protein in peripheral blood leukocytes (PBL). Elevated levels of CD24 may be indicative of colorectal adenoma (inclusive of optically detectable early adenoma to late adenoma, and cancer).

ELIGIBILITY:
Inclusion Criteria:

* Subject is 50 years old and above
* Subject is asymptomatic and referred for regular recommended screening colonoscopy or subject is referred due to suspicion of colon cancer, prior to beginning of any treatment (enriched population)
* Subject signed the informed consent

Exclusion Criteria:

* Subject has been previously diagnosed with any type of cancer
* Subject has been previously diagnosed with a colorectal abnormality such as colorectal adenoma, hyperplastic polyp or carcinoma
* Blood sample was not collected on the day of colonoscopy and prior to colonoscopy
* Subject has first degree family history of colorectal cancer
* Subject has active infection or inflammation as determined clinically at screening
* Subject is currently taking medications related to the previous exclusion criteria
* Subject has participated in, or is participating in, any investigational drug or device study within 30 days prior the date of colonoscopy and any additional study required test
* Pregnant or lactating woman

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects aged 50 years and above that are referred to colonoscopy assessment
Sampling Method: Probability Sample
Enrollment: 229 (Actual)
Dates: Start 2011-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Colonoscopy and CD24 assay correlation | 12 months

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Bat Yamon Gastroentrology Clinic, Bat Yam
  - Zamenhoff Gastroentrology Clinic, Tel Aviv